CLINICAL TRIAL: NCT07107035
Title: Multimodal Large Model-Driven Risk and Prognosis Assessment for Brain Metastases in Lung Cancer: A Nationwide, Multicenter, Observational Study
Brief Title: Multimodal Large Model-Driven Risk and Prognosis Assessment for Brain Metastases in Lung Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhengfei Zhu, Professor, Fudan University
Other Study IDs: LCBM-AI
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: AI (Artificial Intelligence); NSCLC Brain Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Construction of AI models (retrospective cohort)
  Interventions: Other: No Intervention: Observational Cohort
- Validation of AI models (prospective cohort)
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No intervention

SUMMARY:
The goal of this nationwide, multicenter observational study is to develop and externally validate multimodal large models that can (1) predict the risk of brain metastases and (2) estimate long-term prognosis in patients with non-small cell lung cancer (NSCLC).

The main questions it aims to answer are:

* Can a multimodal large model that fuses imaging, pathology, genomic, and clinical data accurately identify NSCLC patients at high risk of developing brain metastases?
* Can a multimodal large model reliably forecast intracranial progression-free survival, progression-free survival, and overall survival across diverse real-world treatment settings? (ie, patients receiving distinct treatment regimens, in different treatment lines and with or without intracranial local therapies).

Because this is an observational study, there are no investigational treatments; instead, researchers will compare outcomes among patients who receive standard-of-care therapies (surgery, radiotherapy, systemic therapy) to determine how well the model's predictions align with observed events.

Participants will:

* Allow use of their routinely collected clinical information, imaging (chest CT, brain MRI), pathology slides, and molecular test results for model training and validation
* Undergo standard-of-care follow-ups
* Complete optional quality-of-life questionnaires during scheduled visits

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years old;
* KPS score≥70;
* Pathologically confirmed lung cancer;
* Receiving guideline-concordant standard-of-care therapy, defined as: radical surgical resection for early- to mid-stage non-small cell lung cancer (NSCLC); stereotactic radiotherapy for early-stage NSCLC deemed medically inoperable; radical chemoradiotherapy for locally advanced NSCLC; or systemic therapy for advanced-stage NSCLC.
* Complete systemic imaging before treatment initiation, including contrast-enhanced brain MRI and contrast-enhanced chest CT;
* Informed consent of the patient.

Exclusion Criteria:

* Multiple primary or metastatic tumors (except early skin cancer, cervical carcinoma in situ that has been treated radically, with no recurrence or progression for more than 5 years);
* Uncontrolled epilepsy, central nervous system disease, or history of mental disorders, judged by the researcher to potentially interfere with the signing of the informed consent form or affect patient compliance;
* Physical examination findings, clinical laboratory abnormalities, or other uncontrolled medical conditions identified by the investigator as potentially interfering with study results interpretation or increasing the patient's risk of treatment complications
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are collected all over China
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
The predictive performance of the multimodal large models | 2 years
  Including Sensitivity (SEN), Specificity (SPE), Matthews Correlation Coefficient (MCC), Area Under the Receiver Operating Characteristic Curve (AUC) with its corresponding 95 % confidence interval (CI)

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 2 years
Intracranial Progression-Free Survival (iPFS) | 2 years
Overall Survival (OS) | 2 years